CLINICAL TRIAL: NCT04697433
Title: Reliability of Myotonometry in Swimming Athletes
Status: Completed | Type: Observational
Sponsor: São Paulo State University (Other)
Responsible Party: Sponsor
Other Study IDs: FIS190047
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Athletes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myotonometry: The evaluation of myotonometry will be carried out by two independent evaluators. The first evaluator will perform the test bilaterally on the middle deltoid, upper trapezius, pectoralis major, biceps brachii, rectus femoris, anterior tibialis, triceps brachii, lumbar multifidus, biceps femoris and soleus previously marked. Immediately after, the second appraiser will perform the same measurements in the same order (Inter-rater reliability). After a 15-minute interval, the retest (intra-rater reliability) will be performed following the same procedure and order as the test step.
  Interventions: Device: Myotonometry

INTERVENTIONS:
Device: Myotonometry — The examiner should exert a slight pressure on the determined point to the necessary depth, which will be indicated by changing the color from red to green light on the device. The device has an automatically controlled preload (0.18 Newton (N)) that will be applied to the contact area by an automatic mechanical pulse, with a duration of 15 milliseconds (ms) and a constant force of 0.4 N , these oscillations will be registered by an accelerometer next to the measurement mechanism inside the device. For each evaluation, a series of 10 consecutive pulses (multiscan mode) will be used with an interval of one second between each pulse. In each shot, the tone, stiffness, elasticity, relaxation time and creep will be calculated.

SUMMARY:
The clinical analysis of athletes has been performed in the sports field to obtain parameters for reliable evaluations. Among the tools used is the myotonometry, an analysis capable of quantitatively measuring tone, stiffness and elasticity. Its reliability has been tested in several populations, however, showing changes in results and presenting high variability in the confidence interval, also, the values of myotonometry differ according to sample specificity and the biomechanical properties of each muscle. Therefore, it seems pertinent to perform the reliability analysis in swimming athletes and verify their applicability and if the values of tone and muscular biomechanical properties vary according to the specificity of the modality. It will be a test and retest study composed of 50 young male and female swimming athletes, aged between 12 and 20 years. The evaluation of myotonometry will be performed randomly by two evaluators and the parameters measured will be: tone, stiffness, elasticity, relaxation time of mechanical stress and displacement. In the test stage, the first evaluator will perform the measurements bilaterally on the muscles and the second evaluator will perform the same measurements in the same order immediately after the first one. After 15 minutes, the retest will be performed following the same order of evaluators in the test. For characterization of sample will be used descriptive statistic through central tendency and variability for all variables collected. Relative reliability will be tested by the Intraclass Correlation Coefficient (ICC). Absolute reliability will be verified by means of standard error of measurement (SEM), values of least detectable change (MMD) and coefficient of variation (CV). The statistical package SPSS Statistics 22.0 will be used to conduct the reliability analyses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy swimming athletes

Exclusion Criteria:

* Being an alcoholic, consuming drugs, smoking or anti-inflammatory and / or analgesic drugs less than 24 hours before the test, presenting anemia, inflammatory process, diabetes, cardiovascular disease, episodes of muscle-tendon or osteoarticular injury in the lower, upper and / or lower limbs spine in the last three months, in addition to swimming for less than two years.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Young swimming athletes who regularly train and are members of the swimming teams of the 4th region of the state of São Paulo, of the São Paulo Aquatic Federation (FAP), of the cities of Presidente Prudente, Votuporanga and São José do Rio Preto.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Muscle Tone | 75 minutes
  MyotonPro (MyotonAS, Tallinn, Estonia), measured in Hertz (Hz)
Stiffness | 75 minutes
  MyotonPro (MyotonAS, Tallinn, Estônia), measured in Newton / meter (N/m)

SECONDARY OUTCOMES:
Elasticity | 75 minutes
  MyotonPro (MyotonAS, Tallinn, Estonia)
Mechanical Stress Relaxation Time | 75 minutes
  MyotonPro (MyotonAS, Tallinn, Estonia), measured in milliseconds (ms)
Creep | 75 minutes
  MyotonPro (MyotonAS, Tallinn, Estonia)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo State, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Individual data will not be disclosed, because as participants are under eighteen